CLINICAL TRIAL: NCT00178854
Title: Risperidone (Risperdal) Augmentation in Depressed Partial Responders to SRI Treatment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: failed recruitment efforts
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030101; RIS-BIP-404; VUMC30141-R; RIS-USA-T31
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
This is a study of the chemistry of depression in people who are taking an antidepressant but it is not working well. The changes in brain chemicals that occur when an SSRI type antidepressant is supplemented with risperidone (Risperdal®) will be studied. Spinal fluid is used to measure chemical levels of dopamine, serotonin, and other chemicals thought to be involved in depression. The study has potential to help understand and treat depression.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-resistant unipolar depression (previous diagnosis of MDD by SCID-P or DSM-IV) as defined by inadequate or waning response to adequate SRI treatment for at least 4 weeks
* HRSD (17-item) score greater than or equal to 15 while taking an SRI with no past suicide attempts for one year and no current ideation, intent, or plan. Repeat HRSD scores should remain greater than or equal to 15 for two consecutive weeks after initial screening.

Exclusion Criteria:

* Adverse extrapyramidal or other response to dopamine antagonist effects in the past.
* Any adverse response to risperidone in the past.
* Residence beyond 30 miles from Vanderbilt University.
* Inability to comply with study requirements.
* Psychotic hallucinations
* Past diagnosis of Bipolar, Dissociative, or Psychotic Disorders.
* Substance or alcohol abuse, other psychotropic, or any investigational or herbal preparation within 3 months or Substance dependency within 6 months prior to initial screening (by SCID-P).
* History of impulsive suicidal gestures or attempts within 2 years (must have no suicidal ideation, intent or plan for a period of one year).
* Primary diagnosis of Cluster B or C personality disorder, or significant comorbidity due to Borderline, Antisocial, Schizoid, or Schizotypal Personality Disorder (by SCID-II).
* Seasonal affective syndromes, including Seasonal Affective Disorder (because the duration of the study is long enough to expect "spontaneous" [natural] remissions.)
* Chronic (daily) benzodiazepine use in the past month or any use 1 week prior to sampling.
* Regular analgesic use. No antipyretic medication is allowed in the pre- through post-sampling period, leaving difficulty with pain management for pain-prone patients.
* Medication use deemed by the investigator unacceptable for study protocol.
* Pregnancy or inability to cooperate with effective contraceptive method (double barrier).
* Physical condition or significant medical history of any illness that presents risk with lumbar catheterization.
* Lactation.
* Blood donation within 90 days prior to or planned 90 days following the study.
* Severe migraine history.
* Daily tobacco use (absolute abstinence is required during the entire study.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2004-05; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Salomon, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States